CLINICAL TRIAL: NCT00960817
Title: "Normal Coronary Artery" With Slow Flow Improved by Adenosine Injection, Dipyridamole Treatment and Clinical Follow-up
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Aaron Frimerman, MD, Hillel Yaffe Medical Center
Other Study IDs: HYMC 02/2009
Record Dates: First submitted 2009-08-17; First posted 2009-08-18 (Estimated); Last update posted 2009-08-18 (Estimated); Status verified 2009-08

CONDITIONS: Coronary Angiography
Keywords: Normal coronary artery with slow blood flow
MeSH Terms: interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; Aspirin; Dipyridamole

ARMS (2):
- 1. Routine treatment (Active Comparator): Control group
  Interventions: Drug: Statin, aspirin
- 2. Dipyridamole treatment (Experimental): Group that receives Dipyridamole treatment
  Interventions: Drug: Dipyridamole

INTERVENTIONS:
Drug: Statin, aspirin
  Arms: 1. Routine treatment
Drug: Dipyridamole
  Arms: 2. Dipyridamole treatment

SUMMARY:
The investigators will investigate patients undergoing coronary angiography with normal coronary but slow blood flow that was normalized after adenosine injection into the coronary artery. The investigators believe that they have small vessel coronary disease which is the initial presentation of coronary disease prior to anatomical narrowing. To alleviate this phenomenon the investigators intend to examine the long-term clinical response of these patients to treatment with dipyridamole, a well-known medication with almost no side-effects that increases the level of adenosine in the tissue.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing coronary angiography and who have normal coronary artery with slow blood flow that normalized with adenosine injection into the coronary artery

Exclusion Criteria:

* Significant coronary disease
* Unstable patients
* Patients with known sensitivity to dipyridamole

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Alleviation of chest pain | Two years

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel